CLINICAL TRIAL: NCT06108687
Title: The Effect of Intraoral Spray Application on Thirst and Thirst Comfort in Patients Undergoing Gynecological Surgery: A Randomized Controlled Study
Brief Title: The Effect of Intraoral Spray Application on Thirst and Thirst Comfort in Patients Undergoing Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zehra Çerçer, Lecturer, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 133
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Application Site Discomfort
Keywords: Gynecologic surgery; water spray; discomfort; thirst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): In cold water applications, 50 cc bottles with plastic spray heads will be used. New materials will be used for each patient. Interventions will be carried out by the researcher and. Cold water kept in the refrigerator at +4 degrees will be placed in 50 cc spray bottles for the experimental group and will be sprayed orally to the patients 3 times an hour in the postoperative period. The spray will be applied to the patient's mouth, upper palate, top of the tongue, right inner cheek, and left inner cheek.
  Patients will be given approximately 0.5 mL of water via spray in each application.
  Interventions: Other: water spray application
- Control (No Intervention): Spray application will not be applied to patients in the control group.

INTERVENTIONS:
Other: water spray application — cold water kept in the refrigerator at +4 degrees
  Arms: Experiment

SUMMARY:
It is important for healthcare professionals to provide care for gynecologic surgery patients using current evidence-based approaches. In this context, this study was planned to determine the effect of intraoral cold water spray application on thirst and thirst comfort in the postoperative period in patients undergoing gynecological surgery.

DETAILED DESCRIPTION:
Hypotheses of the Research H01: Application of cold water spray into the mouth has no effect on thirst in patients undergoing gynecological surgery.

H02: Application of cold water spray into the mouth has no effect on thirst comfort in patients undergoing gynecological surgery.

H11: Application of cold water spray into the mouth has an effect on thirst in patients undergoing gynecological surgery.

H12: Application of cold water spray into the mouth has an effect on thirst comfort in patients undergoing gynecological surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being a patient who is scheduled for benign laparoscopic elective gynecological surgery under general anesthesia,
* No upper gastrointestinal system anomaly and/or disease,
* Being a patient whose score is classified as grade I or II according to the American Society of Anesthesiologists (ASA),
* Being between the ages of 18-65,
* Not smoking,
* Being able to communicate at a level that can answer research questions.

Exclusion Criteria:

* The integrity of the oral and tongue mucosa is disrupted before surgery,
* Having cognitive impairment or any neurological, renal, cardiac or pulmonary chronic disease,
* Morbidly obese
* Those who use psychiatric drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 58 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Thirst Severity Scale (Numerical Rating Scale) | 1st, 3rd, 5th, 6th hours postoperatively
  This scale was determined based on studies in the literature where the severity of thirst was evaluated using a numerical rating scale. It will be used to objectively evaluate the thirst levels of patients. It will be evaluated between 0-10 points with SDQ. While a score of 0 indicates that there is no thirst, a score of 10 indicates that the most severe thirst is felt. (Lee et al. 2020).

SECONDARY OUTCOMES:
Thirst Discomfort Scale | 1st, 3rd, 5th, 6th hours postoperatively
  The Turkish validity and reliability of the scale was conducted by Çiftçi et al. in 2023. The scale is used to determine the level of dehydration-related discomfort in surgical patients. There are 3 sub-dimensions in the scale (intraoral movements, psychological movements, extraoral movements). The scale was developed as a 5-point Likert type. It is scored as "1 = It does not bother me at all", "5 = It bothers me a lot". The Thirst Disorder Scale is calculated based on the total item score. There are no reverse items in the scale. The lowest score from the scale is 12 and the highest score is 60. As the score obtained from the sub-dimension increases, the level of discomfort in that dimension increases. As the score obtained from the scale increases, the level of thirst discomfort of patients increases (Çiftçi et al., 2023).

CONTACTS AND LOCATIONS:
Overall Officials: Zehra ÇERÇER, PhD, Principal Investigator — Gaziantep İslam Science and Technology University; Serap GÜNGÖR, PhD, Study Chair — Kahramanmaras Sutcu Imam University; Esra BULMUŞ, Msc, Study Chair — Adana City Training Hospital; Sefa ARLIER, MD, Study Chair — Adana City Training Hospital
Locations (1):
- Adana city training and research hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oztas M, Oztas B. Effect of Spray Use on Mouth Dryness and Thirst of Patients Undergoing Major Abdominal Surgery: A Randomized Controlled Study. J Perianesth Nurs. 2022 Apr;37(2):214-220. doi: 10.1016/j.jopan.2021.04.018. Epub 2022 Feb 10. PMID 35153118
- [Background] Can S, Gezginci E, Yapici N. Effect of menthol lozenges after extubation on thirst, nausea, physiological parameters, and comfort in cardiovascular surgery patients: A randomized controlled trial. Intensive Crit Care Nurs. 2023 Jun;76:103415. doi: 10.1016/j.iccn.2023.103415. Epub 2023 Feb 20. PMID 36812765
- [Background] Lee CW, Liu ST, Cheng YJ, Chiu CT, Hsu YF, Chao A. Prevalence, risk factors, and optimized management of moderate-to-severe thirst in the post-anesthesia care unit. Sci Rep. 2020 Sep 30;10(1):16183. doi: 10.1038/s41598-020-73235-5. PMID 32999369
- [Background] Ciftci B, Yildiz GN, Avsar G, Kose S, Aydin E, Dogan S, Celik S. Development of the Thirst Discomfort Scale: A Validity and Reliability Study. Am J Crit Care. 2023 May 1;32(3):176-183. doi: 10.4037/ajcc2023954. PMID 37121897